CLINICAL TRIAL: NCT00851669
Title: Behavioral Treatment for Alcohol Dependent Women With Co-occurring Depression
Brief Title: The MEADOW PROJECT (Mending the Effects of Alcohol and Depression on Women) and The Bridge Program (Connecting Recovery Treatment and Behavioral Health)
Acronym: MEADOW/Bridge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Stephanie Gamble, Assistant Professor Department of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00023495; NIH Grant 1K23AA017246-01A1
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Alcohol Dependence; Depression
Keywords: depression; alcohol dependence; women; psychotherapy; men
MeSH Terms: conditions — Alcoholism; Depression; Multiple Endocrine Neoplasia Type 1 | interventions — Interpersonal Psychotherapy; Ethanol; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPT (Experimental): Interpersonal Psychotherapy for Co-occurring Alcohol Dependence and Major Depression (IPT-ADMD) is Interpersonal Psychotherapy with modifications specifically designed for the treatment of patients with co-occurring alcohol dependence and major depression
  Interventions: Behavioral: Interpersonal Psychotherapy for Co-occurring Alcohol Dependence and Major Depression (IPT-ADMD)
- Treatment as Usual (Active Comparator): Individual psychotherapy following usual care practice in a chemical dependency treatment program.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Co-occurring Alcohol Dependence and Major Depression (IPT-ADMD) — Interpersonal Psychotherapy for Co-occurring Alcohol Dependence and Major Depression (IPT-ADMD) is Interpersonal Psychotherapy with modifications specifically designed for the treatment of patients with co-occurring alcohol dependence and major depression
  Arms: IPT
Behavioral: Treatment as Usual — Individual psychotherapy following usual care practice in a chemical dependency treatment program.
  Arms: Treatment as Usual

SUMMARY:
The aim of this study is to evaluate an interpersonally-focused intervention (Interpersonal Psychotherapy) for women with co-occurring alcohol dependence and depression. A sub-protocol has been added to pilot the current study with men with co-occurring alcohol dependence and depression.

DETAILED DESCRIPTION:
Co-occurring alcohol dependence and major depression (AD-MD) is a serious and common public health problem, yet one that is largely unaddressed by conventional chemical dependency treatment. Among alcohol dependent patients, co-occurring depression is associated with poorer treatment outcomes, increased risk for relapse, worse long-term social and functional adjustment, and higher probability of dire outcomes such as suicide. Treatment research on AD-MD patients is needed to inform effective practice. This study provides an initial test of the applicability of Interpersonal Psychotherapy for alcohol dependent women with major depression (IPT-ADMD). The goal of the proposed research project is to refine and test a behavioral intervention that addresses women's co-occurring alcohol dependence and depression within a cohesive interpersonal frame. In Phase 1 of the project, IPT-ADMD will be piloted with 15 AD-MD women enrolled in a MICA (mentally-ill chemical abusers) group treatment program. Findings from Phase 1 will be used to refine the treatment, assessment, and therapist training procedures. In Phase 2, a randomized controlled trial with 60 AD-MD women will be conducted 1) to determine IPT-ADMD's feasibility and acceptability as an adjunct to standard MICA group treatment, and 2) to assess the comparative effects of IPT-ADMD to treatment-as-usual individual therapy (TAU-IT). Compared to TAU-IT, IPT-ADMD is hypothesized to lead to greater reductions in women's drinking frequency, drinking intensity, and depressive symptoms, and to improved interpersonal functioning.

In addition to the current intervention study comparing IPT-ADMD with TAU-IT, we are piloting IPT-ADMD with men in a sub-protocol of the main study. The target population of the Bridge Program will be men with alcohol dependence and co-occurring major depression. We hypothesize that IPT will be feasible and acceptable and will improve drinking frequency and intensity; depressive symptoms; and interpersonal functioning. The proposed sub-protocol will allow us to determine if future clinical trials of IPT should include both male and female patients with co-occurring alcohol dependence and depression.

ELIGIBILITY:
Inclusion Criteria:

* Current Alcohol Dependence and Major Depression

Exclusion Criteria:

* Bipolar Disorder
* Psychosis or schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-back Interview (percentage days abstinent, average drinks per drinking day) | Baseline, 8 weeks, 16 weeks, 24 weeks, and 32 weeks for women; Baseline, 8 weeks, and 16 weeks for men

SECONDARY OUTCOMES:
Beck Depression Inventory | Baseline, 8 weeks, 16 weeks, 24 weeks, and 32 weeks for women; Baseline, 8 weeks, and 16 weeks for men
Hamilton Rating Scale for Depression | Baseline, 8 weeks, 16 weeks, 24 weeks, and 32 weeks for women; Baseline, 8 weeks, and 16 weeks for men

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Gamble, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States